CLINICAL TRIAL: NCT07128485
Title: Remote Fentanyl Test Strip Distribution and Education to Prevent Drug Overdose
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Emma Kay, Associate Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB 300015053
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Accidental Overdose of Opiate
Keywords: overdose prevention; fentanyl test strips; fentanyl; opioid use disorder; stimulant use disorder; accidental overdose
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Using a 2x2 design, there will be four study arms. All arms will be given a resource list on where to obtain naloxone and fentanyl test strips (FTS), while other arms will additionally receive mail-distributed FTS, FTS education, or both. These 4 groups include: FTS distribution + education (FDE), FTS education (E), FTS distribution only (FD), and a control group (referral only).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FDE (Experimental): This arm receives both FTS distribution (FTS delivered to their residential address) and education (FDE), as well as a resource list for naloxone and additional FTS if desired.
  Interventions: Other: Fentanyl test strips; Behavioral: Fentanyl test strip education
- E (Experimental): The Education only (E) arm receives FTS education as well as a resource list for obtaining naloxone and FTS.
  Interventions: Behavioral: Fentanyl test strip education
- FD (Experimental): The FTS distribution only (FDE) arm receives FTS delivered to their residential address as well as a resource list for obtaining naloxone and additional FTS, if desired.
  Interventions: Other: Fentanyl test strips
- R (No Intervention): The referral only (R) arm receives a resource list for obtaining naloxone and FTS.

INTERVENTIONS:
Other: Fentanyl test strips — Fentanyl test strips (FTS) are small strips of paper that can detect the presence of fentanyl in illicit drugs.
  Arms: FD; FDE
Behavioral: Fentanyl test strip education — Developed in the R61 phase, the educational intervention will provide participants with knowledge about how to correctly use fentanyl strips.
  Arms: E; FDE

SUMMARY:
This Type 1 hybrid effectiveness-implementation randomized controlled trial, Remote Fentanyl Test Strip Distribution and Education to Prevent Drug Overdose, aims to address the United States opioid crisis driven by fentanyl and other synthetic opioids by reducing overdose rates. This study would be the first national, fully remote trial to assess the impact of fentanyl test strips on overdose outcomes, using a novel 2x2 design crossing fentanyl test strip distribution and education to determine which approach most significantly reduces overdose rates while minimizing costs. This research will inform scalability around mail-based fentanyl test strip distribution and education programs to address the nation's opioid overdose crisis.

DETAILED DESCRIPTION:
This Type 1 hybrid effectiveness-implementation randomized controlled trial, Remote Fentanyl Test Strip Distribution and Education to Prevent Drug Overdose, aims to address the United States opioid crisis driven by fentanyl and other synthetic opioids. Fentanyl test strips (FTS) are a cheap, low burden tool used to detect the presence of fentanyl in drugs, and they are associated with high acceptability, yet critical FTS knowledge and implementation gaps persist. Moreover, extant studies of FTS programs are either limited to one city or region and enroll from brick-and-mortar sites, with no remote randomized controlled trials (RCTs) to date. This study would be the first national, fully remote RCT to assess the impact of FTS on overdose outcomes among people using illicit stimulants and/or opioids. This project adapts the investigators' Remote Opioid Overdose Education and Naloxone Distribution intervention to FTS using a human-centered design approach, leveraging partnerships with national and regional community partners to co-create a fully remote intervention.

The study will use a 2x2 design to cross remote FTS distribution with remote FTS education, thereby isolating the individual and combined effects of the two components. The R61 phase focuses on adapting and piloting the interventions with 100 participants, assessing feasibility, acceptability, and appropriateness. The R33 phase implements a fully powered trial to compare overdose outcomes (fatal and non-fatal) among 2,952 participants randomized to the four study arms, which include: FTS distribution and education, FTS education only, FTS distribution only, and a control group. All groups will receive a resource list for naloxone and FTS. The secondary outcome is FTS knowledge, while exploratory outcomes include behavioral strategies to reduce risk of overdose (including FTS-specific behaviors) and utilization of substance use services engagement and treatment. The study also incorporates ecological momentary assessment to offer insights into daily contextual factors influencing FTS use, as well as a cost-effectiveness analysis to determine the most cost-effective approach with most overdoses averted. The study's 2x2 design allows for a thorough examination of the interactions between FTS distribution and education, identifying the most effective and cost-efficient approach for reducing overdose rates. Overall, findings will inform the scalability of remote overdose prevention interventions. This work represents a sustainable, fully remote model that can be implemented nationwide, setting the stage for transformative advancements in overdose prevention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* English-speaking and reading
* Report using illicit opioids and/or stimulants (including counterfeit pills) within the past 3 months per the ASSIST
* Able and willing to provide informed consent
* Reside in any of the US states where fentanyl test strips are legal with no plans to move out of state for at least 12 months
* Reside in any of the US states where FTS are legal with no plans to move out of state for at least 12 months
* Be able and willing to provide the names and contact information of three close contacts to reach if the participant cannot be reached

Exclusion Criteria:

* Living in a restricted environment (e.g., prison)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Overdose | Baseline, 1 month, 3 months, 6 months
  Includes both self-reported non-fatal overdose and fatal overdose as reported by the National Death Index.

SECONDARY OUTCOMES:
Fentanyl test strip knowledge | Baseline, 1 month, 3 months, 6 months
  Self-reported knowledge of how and when to use fentanyl test strips correctly, based on the fentanyl test strip education intervention developed in R61 phase

OTHER OUTCOMES:
Protective Behavioral Strategies | Baseline, 1 month, 3 months, 6 months
  Self-reported behavioral strategies to reduce risk of opioid overdose, based on an 8-item composite measure.
Types of drugs tested with fentanyl test strips | Baseline, 1 month, 3 months, 6 months
  Self-reported list of all types of drugs tested with fentanyl test strips
Number of fentanyl test strips used | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months
  Self-reported number of fentanyl test strips used over reporting period
Results of fentanyl test strips | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months
  Self-report of number of fentanyl test strips that tested positive, negative, and unclear or invalid results during reporting period
Substance Use Service Engagement and Treatment | Baseline, 1 month, 3 months, 6 months
  Self-report measure of participants' use of other substance use related services not measured elsewhere (e.g., intensive outpatient programs, residential treatment)
Fentanyl test strip referral accessibility | Baseline, 1 month, 3 months, 6 months
  Self report of ease of obtaining fentanyl test strips from referral sources provided in the study and which referral sources were accessed

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No